CLINICAL TRIAL: NCT06179641
Title: Analgesic Efficacy of IPACK Versus Selective Tibial Nerve Block in Patients Undergoing Total Knee Arthroplasty Under Spinal Anesthesia With an Adductor Canal Block: a Randomized Controlled Double-blinded Trial
Brief Title: Comparison of Two Different Regional Analgesia Techniques for Patients Undergoing Total Knee Arthroplasty
Acronym: PIPACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Prof. Dr. Med. Eric Albrecht, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-VD 2023-02041
Record Dates: First submitted 2023-11-30; First posted 2023-12-22 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Analgesia; Arthropathy of Knee; Postoperative Pain
Keywords: nerve block; pain management; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: single centered, prospective, randomized double blinded controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPACK group (Active Comparator): IPACK (Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee) block
  Interventions: Procedure: IPACK block
- Tibial nerve group (Experimental): selective tibial nerve block
  Interventions: Procedure: Selective tibial nerve block

INTERVENTIONS:
Procedure: Selective tibial nerve block — The selective tibial nerve block will be performed on the popliteal crease following sterilization of the area. The probe will be placed in a transverse position at the popliteal crease to visualize the popliteal artery and the tibial nerve in short axis. A 21-gauge 50mm insulated facet tip needle (SonoPlex® STIM, Pajunk, Geisingen, DE) will be inserted in-plane with the ultrasound bean from a medial to lateral direction. Once the needle tip is adjacent to the tibial nerve, 5 ml of ropivacaine 0.75% will be injected to achieve an adequate spread of local anesthetics around the nerve.
  Arms: Tibial nerve group
Procedure: IPACK block — The IPACK (Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee) will be performed on the popliteal crease following sterilization of the area. The probe will be placed in a transverse position proximal to the popliteal crease to visualize the popliteal artery in short axis. A 21-gauge 100 mm insulated facet tip needle (SonoPlex® STIM, Pajunk, Geisingen, DE) will be inserted in-plane with the ultrasound beam, in a lateral to medial direction, between the popliteal artery and the posterior capsule, where nineteen mL of ropivacaine 0.2% will be injected under ultrasound guidance. The distribution of local anesthetics will be observed above the posterior capsule.
  Arms: IPACK group

SUMMARY:
The objective of this clinical trial is to compare two regional analgesia techniques in patients undergoing total knee arthroplasty: IPACK (Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee) vs selective tibial nerve block. The main question is whether one of these peripheral blocks is more effective in reducing postoperative pain than the other. All patients will have a spinal block with an adductor canal block. One group will receive an IPACK block and the other group, a selective tibial nerve block. Postoperative pain scores and morphine consumption, among others, will be compared between groups.

DETAILED DESCRIPTION:
The aim of this randomized controlled double blinded trail is to compare an analgesic effect of an IPACK (Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee) block vs selective tibial nerve block in patients scheduled for total knee arthroplasty under spinal anesthesia with an adductor canal block.

The investigators presume that association of a selective tibial nerve block with an adductor canal block provides better postoperative analgesia than a combination of an IPACK (Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee) block with an adductor canal block. The research team plan on including 100 patients and randomly assign them to two groups of 50 patients each. After written informed consent, patients will be allocated to one of the groups, following a computer-generated list of randomization. All patients will receive central spinal anesthesia with 12.5 mg of hyperbaric bupivacaine with 100 mcg of morphine and an adductor canal block with 150 mg of ropivacaine. IPACK block group will then receive an IPACK block with 38 mg of ropivacaine and a tibial nerve group will receive a selective tibial nerve block with 37.5 mg of ropivacaine.

During the surgery, iv dexamethasone 8 mg, iv magnesium sulfate 40 mg.kg-1, iv ketorolac 30 mg, and iv acetaminophen 1000 mg. will be administered to all patients.

After surgery, all patients will be prescribed an iv patient-controlled analgesia (PCA) of morphine (boluses of 2 mg available every 10 min, maximum of 40 mg every 4 hours) along with oral acetaminophen (1000 mg every 6 h) and oral ibuprofen (400 mg every 8 hours). Oral ondansetron 4 mg every 8 hours will be available on request in case of nausea or vomiting.

The primary outcome will be the cumulative iv morphine consumption at 24 h postoperatively. Secondary outcomes will include pain- and functional-related outcomes. Pain related outcomes are cumulative morphine consumption in the recovery room, at day 1, day 2 and day 3 postoperatively, rest and dynamic pain scores, duration of peripheral nerve block defined as the time between the execution of the block and the first dose of iv morphine, incidence of postoperative nausea and vomiting and pruritus during 3 days following surgical intervention, incidence of peroneal nerve block and complications of peripheral nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification I-III
* 18 yo or older
* patients scheduled for total knee arthroplasty under central spinal anesthesia
* informed consent signed

Exclusion Criteria:

* Refusal or inability for informed consent
* Known allergies to ropivacaine, acetaminophen, ibuprofen, ketorolac, morphine, ondansetron or dexamethasone
* Secondary surgical revision
* Opioid treatment such as morphine, hydrocodone, hydromorphone, tramadol, methadone, fentanyl, buprenorphine or codeine
* Bleeding diathesis
* Neurological deficit
* Known renal insufficiency (eGFR <45 ml/min)
* Known hepatic insufficiency (Child score B or C)
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
Total iv morphine consumption | 24 hours postoperatively
  consumption in mg

SECONDARY OUTCOMES:
Morphine consumption in the recovery room | From admission till discharge from the recovery room, up to 2 hours
  consumption in mg
PCA administered morphine consumption | at day 1, day 2 and day 3 postoperatively
  consumption in mg administered by PCA
rest and dynamic pain scores | at day 1, day 2 and day 3 postoperatively
  Visual Analogue scale(VAS), 0-10 where 0 is no pain and 10 is the worst pain imaginable
Duration of peripheral nerve block | From execution of a peripheral nerve block till administration of a first dose of iv morphine, up to 48 hours
  Time between execution of a peripheral nerve block and the first dose of iv morphine
Incidence of postoperative nausea and vomiting | at day 1, day 2 and day 3 postoperatively
  Presence of nausea and vomiting in the postoperative period
Incidence of pruritus | at day 1, day 2 and day 3 postoperatively
  Presence of pruritus
peroneal nerve block | at day 1, day 2 and day 3 postoperatively
  presence of peroneal nerve block
complications of peripheral nerve blocks | at the moment of execution of the block (day 0) and at day 3 postoperatively
  iv injection, hematoma, infection
passive and active motion range | at day 3 postoperatively
  joint motion in degrees
quadriceps strength | at day 3 postoperatively
  Percentage of strength as compared with the opposite leg
walking distance | at 72h postoperatively
  walking distance without pain
hospital stay | from admission to the hospital till discharge, up to 3 days
  length of hospital stay in days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] Williams DP, O'Brien S, Doran E, Price AJ, Beard DJ, Murray DW, Beverland DE. Early postoperative predictors of satisfaction following total knee arthroplasty. Knee. 2013 Dec;20(6):442-6. doi: 10.1016/j.knee.2013.05.011. Epub 2013 Jun 16. PMID 23777807
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] van der Wal M, Lang SA, Yip RW. Transsartorial approach for saphenous nerve block. Can J Anaesth. 1993 Jun;40(6):542-6. doi: 10.1007/BF03009739. PMID 8403121
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Silverman ER, Vydyanathan A, Gritsenko K, Shaparin N, Singh N, Downie SA, Kosharskyy B. The Anatomic Relationship of the Tibial Nerve to the Common Peroneal Nerve in the Popliteal Fossa: Implications for Selective Tibial Nerve Block in Total Knee Arthroplasty. Pain Res Manag. 2017;2017:7250181. doi: 10.1155/2017/7250181. Epub 2017 Feb 2. PMID 28260964
- [Background] Paulou F, Wegrzyn J, Rossel JB, Gonvers E, Antoniadis A, Kagi M, Wolmarans MR, Lambert J, Albrecht E. Analgesic efficacy of selective tibial nerve block versus partial local infiltration analgesia for posterior pain after total knee arthroplasty: a randomized, controlled, triple-blinded trial. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101223. doi: 10.1016/j.accpm.2023.101223. Epub 2023 Apr 6. PMID 37030393